CLINICAL TRIAL: NCT05501561
Title: A Phase 2b, Randomized, Observer-Blind, Antigen and Adjuvant Dose-Confirmation Clinical Study to Evaluate Safety and Immunogenicity of Different Formulations of MF59-Adjuvanted Quadrivalent Subunit Inactivated Cell-derived Influenza Vaccine (aQIVc) in Older Adults ≥50 Years of Age
Brief Title: Safety and Immunogenicity of Different Formulations of an MF59-Adjuvanted Influenza Vaccine in Older Adults ≥50 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V201_07
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Influenza, Human
Keywords: influenza, vaccine, MF59, adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IIV-A Investigational (Experimental)
  Interventions: Biological: Experimental: IIV-A Investigational IIV-A will be administered as a single dose intramuscularly on Day 1
- aIIV-B Investigational (Experimental)
  Interventions: Biological: Experimental: aIIV-B Investigational aIIV-B will be administered as a single dose intramuscularly on Day 1
- aIIV-C Investigational (Experimental)
  Interventions: Biological: Experimental: aIIV-C Investigational aIIV-C will be administered as a single dose intramuscularly on Day 1
- Licensed IIV (Active Comparator)
  Interventions: Biological: Active Comparator: Licensed IIV IIV will be administered as a single dose intramuscularly on Day 1

INTERVENTIONS:
Biological: Experimental: IIV-A Investigational IIV-A will be administered as a single dose intramuscularly on Day 1 — Biological/Vaccine: Investigational IIV-A Investigational Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: IIV-A Investigational
Biological: Experimental: aIIV-B Investigational aIIV-B will be administered as a single dose intramuscularly on Day 1 — Biological/Vaccine: Investigational aIIV-B Investigational MF59 Adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: aIIV-B Investigational
Biological: Experimental: aIIV-C Investigational aIIV-C will be administered as a single dose intramuscularly on Day 1 — Biological/Vaccine: Investigational aIIV-C Investigational MF59 Adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: aIIV-C Investigational
Biological: Active Comparator: Licensed IIV IIV will be administered as a single dose intramuscularly on Day 1 — Biological/Vaccine: Licensed IIV Licensed Non-adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Licensed IIV

SUMMARY:
This Phase 2, randomized, observer-blind, dose-confirmation Clinical study is evaluating different formulations of MF59-Adjuvanted Quadrivalent Subunit Inactivated Influenza Vaccine. Approximately 1000 subjects are to be randomized into 1 of 4 possible treatment groups with 250 participants per group. Every participant will receive an influenza vaccine injection on Day 1 and will be followed up for approximately 6 months following injection. The primary immunogenicity analysis is based on Day 29 serology data.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, all subjects must meet ALL of the inclusion criteria described.

1. Individuals ≥50 years of age on the day of informed consent.
2. Individuals who have voluntarily given written consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Individuals who can comply with study procedures including follow-up .
4. Males, females of non-childbearing potential or females of childbearing potential who are using an effective birth control method, at least 30 days prior to informed consent, which they intend to use for at least 2 months after the study vaccination.

   -

Exclusion Criteria:

In order to participate in this study, all subjects must not meet ANY of the exclusion criteria described below:

1. Females of childbearing potential who are pregnant, lactating, or who have not adhered to a specified set of contraceptive methods from at least 30 days prior to informed consent and who do not plan to do so for at least 2 months after the study vaccination.
2. Progressive, unstable or uncontrolled clinical conditions.
3. Hypersensitivity, including allergy, to any component of vaccines whose use is foreseen in this study.
4. History of any medical condition considered an adverse event of special interest (AESI).
5. Known history of Guillain-Barré syndrome or another demyelinating disease such as encephalomyelitis and transverse myelitis.
6. Clinical conditions representing a contraindication to intramuscular administration of vaccines or blood draw.
7. Abnormal function of the immune system resulting from:

   1. Clinical conditions.
   2. Systemic administration of corticosteroids (PO/IV/IM) at a dose of ≥20 mg/day of prednisone or equivalent for more than 14 consecutive days within 90 days prior to informed consent5.
   3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
8. Receipt of immunoglobulins or any blood products within 180 days prior to informed consent.
9. Receipt of an investigational or non-registered medicinal product within 30 days prior to informed consent.
10. Receipt of any COVID-19 vaccine within 14 days (non-replicating vaccines) or 28 days (replicating vaccines) prior to informed consent or plan to receive any COVID-19 vaccine within 7 days from study vaccination
11. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to informed consent or who are planning to receive any vaccine within 28 days from the study vaccines.
12. Study personnel or immediate family or household member of study personnel.
13. Receipt of any influenza vaccine within 6 months prior to informed consent, or plan to receive an influenza vaccine during the study period.
14. Acute (severe) febrile illness,
15. Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.

    -

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1056 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Immunogenicity Endpoint: Hemagglutination inhibition (HI) titers against vaccine A and B influenza strains | 28 days post-vaccination
The Percentage of Subjects with Solicited Local and Systemic Reactions | 7 days post-vaccination
The Percentage of Subjects with Unsolicited Adverse Events | 28 days post-vaccination
The Percentage of Subjects with Serious Adverse Events (SAEs), AEs Leading to Withdrawal, Adverse Events of Special Interest (AESI) and Medically Attended Adverse Events (MAAEs) | 180 days post-vaccination

SECONDARY OUTCOMES:
Immunogenicity Endpoint: Microneutralization (MN) titers against vaccine A and B influenza strains | 28 days post-vaccination

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - AMR Tempe, Tempe, Arizona
  - Marvel Clinical Research, Huntington Beach, California
  - California Research Center, San Diego, California
  - The Lynn Institute of The Rockies, Colorado Springs, Colorado
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Velocity Clinical Research - New Smyrna Beach, Edgewater, Florida
  - CenExel RCA, Hollywood, Florida
  - Health Awareness INC, Jupiter, Florida
  - Global Health Research Center, Miami Lakes, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Global Health Research Center, Tampa, Florida
  - Platinum Research Network, LLC, Savannah, Georgia
  - Meridian Clinical Research - Savannah, Savannah, Georgia
  - AMR El Dorado, El Dorado, Kansas
  - AMR Lexington, Lexington, Kentucky
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - Medpharmics, LLC, Metairie, Louisiana
  - Rockville Internal Medicine Group, Rockville, Maryland
  - MedPharmics LLC, Biloxi, Mississippi
  - Healthcare Research Network, Hazelwood, Missouri
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research, Bellevue, Nebraska
  - Meridian Clinical Research, Grand Island, Nebraska
  - Meridian Clinical Research, LLC, Lincoln, Nebraska
  - Alliance for Multispecialty Research, LLC, Las Vegas, Las Vegas, Nevada
  - Meridian Clinical Research (Binghamton, NY), Binghamton, New York
  - Meridian Clinical Research, LLC, Endwell, New York
  - Velocity Clinical Research - Syracuse, Syracuse, New York
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Aventiv Research, Inc. Columbus, Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Velocity Clinical Research, Gaffney, Gaffney, South Carolina
  - Velocity Clinical Research - Greenville, Greenville, South Carolina
  - Velocity Clinical Research, Spartanburg, Spartanburg, South Carolina
  - Meridian Clinical Research - Dakota Dunes, Dakota Dunes, South Dakota
  - AMR Coastal Clinical Research, Knoxville, Tennessee
  - DM Clinical Research, Tomball, Texas
  - JBR Clinical Research, Salt Lake City, Utah
  - Velocity Clinical Research - West Jordan, West Jordan, Utah
  - CVS pharmacy - Charlottesville, Charlottesville, Virginia
  - CVS pharmacy - Reston, Reston, Virginia
  - CVS pharmacy - Richmond, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
SEQIRUS supports the release of anonymized subject-level and study-level data in compliance with regulatory requirements, including Clinical Documents which are part of the CTD modules submitted to regulatory agencies for public release.
  Summary results disclosure is either in document form (e.g., ICH E3 Clinical Study Report synopsis) or structured data form (such as summary results in ClinicalTrials.gov (United States) or eudract.ema.europa.eu (EU Clinical Trial Registry [EU CTR])
Supporting Information: Study Protocol, SAP
Time Frame: SEQIRUS discloses results from clinical studies within 12 months of completion of the study unless otherwise mandated by local laws or regulations.
Access Criteria: SEQIRUS will consider requests from qualified scientific and medical researchers to disclose protocols, anonymized subject-level data and study-level data when there is medical, scientific and/or public health interest to ensure the safe use of a Seqirus product licensed on or after 1 January 2014 in the United States (US) and/or the European Union (EU). This applies to Seqirus-sponsored interventional studies initiated after 27 September 2007 and ongoing as of 26 December 2007, that have been included as part of a US or EU submission package which received approval in US and EU on or after 1 January 2014 and have been accepted for publication
URL: http://www.seqirus.us/partnering